CLINICAL TRIAL: NCT05280574
Title: Continuous Ward Monitoring With the GE Portrait Mobile Monitoring Solution: the COSMOS Trial A Pilot Study
Brief Title: The COSMOS Trial. A Pilot Study A Pilot Study
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 21-970
Record Dates: First submitted 2022-02-22; First posted 2022-03-15 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Phase 1 - prospective observational cohort study: Blinded GE Portrait monitoring: Patients in phase 1 will receive continuous vital sign monitoring blinded to patients and clinicians.
  Interventions: Device: Blinded GE Portrait Monitoring
- Phase 2- randomized trial: Blinded GE Portrait monitoring: Continuous vital signs will be monitored and recorded in patients assigned to blinded monitoring, but were not available to clinicians, who instead will rely on routine vital sign assessments at 4-hour intervals.
  Interventions: Device: Blinded GE Portrait Monitoring
- Phase 2- randomized trial: Unblinded GE Portrait monitoring: Physician investigators will monitor and evaluate continuous vital sign data 24 hours per day for patients assigned to unblinded GE Portrait monitoring. Patients who are randomized to the unblinded GE Portrait monitoring might be intervened if the clinicians believe that the alarm is clinically meaningful.
  Interventions: Device: Unblinded GE Portrait Monitoring

INTERVENTIONS:
Device: Blinded GE Portrait Monitoring — Continuous vital signs will be monitored and recorded by GE Portrait but not available to clinicians.
  Groups: Phase 1 - prospective observational cohort study: Blinded GE Portrait monitoring; Phase 2- randomized trial: Blinded GE Portrait monitoring
Device: Unblinded GE Portrait Monitoring — Continuous vital signs will be monitored and evaluated by clinicians using GE Portrait.
  Groups: Phase 2- randomized trial: Unblinded GE Portrait monitoring

SUMMARY:
The investigators plan a pilot study to evaluate patient tolerance of the GE Portrait Mobile Monitoring Solution, along with appropriate alert thresholds, and clinical utility. Data obtained in the proposed pilot cohort will guide design of a future robust randomized trial comparing clinical interventions and serious complications with blinded versus unblinded continuous ward monitoring.

DETAILED DESCRIPTION:
The investigators plan a pilot study to evaluate patient tolerance of the GE Portrait Mobile Monitoring Solution, along with appropriate alert thresholds, and clinical utility. The system is a novel battery-powered untethered monitor for continuous monitoring of oxygen saturation, respiratory rate, and pulse rate that is designed for use by patients on surgical wards. The initial phase will evaluate patient tolerance, with clinicians and patients blinded to monitor data. Results will be used to evaluate the frequency of respiratory events and pulse rate abnormalities. These data will be used to design clinical alert settings, based on various durations at various thresholds (e.g., saturation <85% for >1 minute). Our main goal will be to identify clinically meaningful vital sign abnormalities with a minimum of false alerts. Secondarily, the investigators will evaluate the frequency and duration of abnormalities, and the fraction that are detected clinically.

In the second phase of the pilot, clinicians will be unblinded to the GE Portrait monitors, and alerts provided based on the durations and threshold identified in the initial part of the pilot. The primary outcomes will be clinician tolerance and the extent to which clinicians believe that vital sign trending and alerts provided useful information rather than distraction. Specifically, the investigators will assess the fraction of alerts that clinicians deemed meaningful, and the fraction that resulted in clinical interventions. In the third phase of the pilot, the durations and thresholds for saturation, respiratory rate, and pulse rate that trigger alerts will be adjusted based on results from the second phase.

ELIGIBILITY:
Inclusion Criteria:

* Are admitted to one of the wards equipped with the GE Portrait Mobile Solution.
* Are designated American Society of Anesthesiologists physical status 1-4.
* Had major noncardiac surgery lasting at least 1.5 hours.
* Are expected to remain hospitalized at least two postoperative nights.
* Had general anesthesia with or without neuraxial anesthesia.

Exclusion Criteria:

* Have language, vision, or hearing impairments that may compromise continuous monitoring.
* Are designated Do Not Resuscitate, hospice, or receiving end of life care
* Have previously participated in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are older than 18 years of age. Patients have a ASA status 1-4. The patients whom had a major noncardiac surgery lasting at least 1.5 hours and are expected to remain hospitalized at least two postoperative nights, and are being admitted to a ward equipped with the GE Portrait Mobile Monitor.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sessler, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Anusic N, Gulluoglu A, Ekrami E, Mascha EJ, Li S, Coffeng R, Turan A, Clemens A, Perez C, Beard JW, Sessler DI; COSMOS Pilot Investigators. Corrigendum to 'Continuous Vital Sign Monitoring on Surgical Wards: The COSMOS Pilot. J Clin Anesth. 2026 Jan;108:111878. doi: 10.1016/j.jclinane.2025.111878. Epub 2025 Oct 30. PMID 41168018
- [Derived] Anusic N, Gulluoglu A, Ekrami E, Mascha EJ, Li S, Coffeng R, Turan A, Clemens A, Perez C, Beard JW, Sessler DI; COSMOS Pilot Investigators. Continuous vital sign monitoring on surgical wards: The COSMOS pilot. J Clin Anesth. 2024 Dec;99:111661. doi: 10.1016/j.jclinane.2024.111661. Epub 2024 Nov 11. PMID 39531997

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 1 enrolled 100 patients with continuous vital sign monitoring blinded to patients and clinicians.
  Phase 2 randomized 150 patients to either blinded or unblinded continuous monitoring.
Pre-assignment Details: Phase 1: A prospective observation cohort phase (no randomization) designed to identify suitable alert thresholds for continuous oxygen saturation, heart rate, and respiratory rate for phase 2. Patient characteristics weren't collected per protocol, ,and analysis was completely qualitative.
  Phase 2: A randomized trial phase. 176 patients consented, 26 patients withdrew before randomization:
  * 21 patients went to ICU after surgery
  * 5 patients declined to attend the study.
Groups:
- Phase 1 - Prospective Observational Cohort Study: Blinded GE Portrait Monitoring: Patients received continuous vital sign monitoring blinded to patients and clinicians.
  Phase 1 was a prospective cohort study without randomization. Patient characteristics weren't collected per protocol, and analysis was completely qualitative.
- Phase 2 - Randomized Trial: Unblinded GE Portrait Monitoring: Physician investigators monitored and evaluated continuous vital sign data 24 hours per day for patients assigned to unblinded GE Portrait monitoring.
- Phase 2 - Randomized Trial: Blinded GE Portrait Monitoring: Continuous vital signs were monitored and recorded in patients assigned to blinded monitoring, but were not available to clinicians, who instead relied on routine vital sign assessments at 4-hour intervals.
Period: Overall Study
Arm/Group | Phase 1 - Prospective Observational Cohort Study: Blinded GE Portrait Monitoring | Phase 2 - Randomized Trial: Unblinded GE Portrait Monitoring | Phase 2 - Randomized Trial: Blinded GE Portrait Monitoring
Started | 100 | 75 | 75
Completed | 100 | 73 | 75
Not Completed | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 2- Randomized Trial: Blinded GE Portrait Monitoring: Continuous vital signs were monitored and recorded in patients assigned to blinded monitoring, but were not available to clinicians, who instead relied on routine vital sign assessments at 4-hour intervals.
- Phase 2- Randomized Trial: Unblinded GE Portrait Monitoring: Physician investigators monitored and evaluated continuous vital sign data 24 hours per day for patients assigned to unblinded GE Portrait monitoring. Patients who are randomized to the unblinded GE Portrait monitoring might be intervened if the clinicians believe that the alarm is clinically meaningful.
- Total: Total of all reporting groups
Arm/Group | Phase 2- Randomized Trial: Blinded GE Portrait Monitoring | Phase 2- Randomized Trial: Unblinded GE Portrait Monitoring | Total
Number analyzed (Participants) | 75 | 73 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (16) | 60 (14) | 59 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 41 | 83
  Male | 33 | 32 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Missing data points: 1 for unblinded group and 2 for blinded group
  Participants
    number analyzed (Participants) | 73 | 72 | 145
    White | 62 | 61 | 123
    Black | 9 | 8 | 17
    Other | 2 | 3 | 5
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Missing data point: 1 for blinded group.
  kg/m^2
    number analyzed (Participants) | 74 | 73 | 147
    (all) | 28 (7.6) | 28 (6.2) | 28 (7.1)
American Society of Anesthesiologists (ASA) physical status [Count of Participants; unit: Participants]
  Normal | 1 | 0 | 1
  Mild | 11 | 10 | 21
  Moderate | 62 | 60 | 122
  Severe | 1 | 3 | 4
Smoking status [Count of Participants; unit: Participants] — Population: Missing data point: 5 for blinded group and 3 for unblinded group
  Participants
    number analyzed (Participants) | 70 | 70 | 140
    Never | 46 | 39 | 85
    Current | 8 | 9 | 17
    Former (> 6 weeks) | 16 | 22 | 38

OUTCOME MEASURES:

1. Primary Outcome: Phase 2- Cumulative Duration of Vital Sign Abnormalities
Description: The vital sign abnormalities is a 5-component composite including the durations of SpO2 <85%, heart rate <45/min, heart rate >130/min, respiratory rate <4/min and respiratory rate >30/min.
Time Frame: Up to 72 hours after surgery
Population: Monitor data for one patient in the blinded group was lost so we assumed that AET for all five outcomes were zero.
Measure: Median (Inter-Quartile Range); unit: minutes beyond threshold
Groups:
- Phase 2- Unblinded GE Portrait Monitoring: Physician investigators will monitor and evaluate continuous vital sign data 24 hours per day for patients assigned to unblinded GE Portrait monitoring.
- Phase 2- Blinded GE Portrait Monitoring: Continuous vital signs will be monitored and recorded in patients assigned to blinded monitoring, but were not available to clinicians, who instead will rely on routine vital sign assessments at 4-hour intervals.
Arm/Group | Phase 2- Unblinded GE Portrait Monitoring | Phase 2- Blinded GE Portrait Monitoring
Number analyzed (Participants) | 73 | 75
minutes beyond threshold
  SPO2 < 85% | 6.2 [1.1 to 17] | 4.2 [0.75 to 37]
  Respiratory rate < 4 breaths/min | 0 [0 to 0] | 0 [0 to 0]
  Respiratory rate > 30 breaths/min | 8.4 [2.3 to 21] | 10 [2.4 to 20]
  Heart rate < 45 beats/min | 0.02 [0 to 1.1] | 0.42 [0 to 2]
  Heart rate > 130 beats/min | 0 [0 to 1.2] | 0 [0 to 0.83]
Statistical Analysis 1: Comparison: Phase 2- Unblinded GE Portrait Monitoring vs Phase 2- Blinded GE Portrait Monitoring; Test type: Other; p < 0.05, Distinct-effects GEE model; Ratio of geometric means = 0.75, 95% CI 2-sided [0.51 to 1.1] — Average relative effect of unblinded versus blinded monitoring across the 5-component composite (SpO2 <85%, RR >30/min, RR <4/min, HR <45/min, HR >130/min) of cumulative durations; We assessed the treatment effect of unblinded versus blinded monitoring across the 5-component primary outcome composite of cumulative durations by estimating the average relative effect on the log-transformed count data (counts of observations beyond a given threshold at 1 Hz). Specifically, we employed a distinct-effects (i.e., separate treatment effect estimated for each component) generalized estimating equation (GEE) model to account for within-subject correlation across components with the vector of the 5 cumulative durations as the dependent variable and treatment as independent. We then averaged the component-specific effects and tested whether the average effect equals zero (on the log scale), and reported results as the ratio of geometric means of unblinded versus blinded monitoring

2. Secondary Outcome: Phase 2 - Alerts Deemed Meaningful
Description: Fraction of alerts deemed as meaningful by clinicians/total alerts in unblinded group
Time Frame: During postoperative 72 hours
Population: We analyzed 73 patients in the unblinded GE Portrait monitoring group, with a total of 73 alarms recorded. Among them, 41 patients experienced no alarms, while the remaining 32 patients accounted for all 73 alarms.
Measure: Number; unit: Meaningful alarms
Units Other Than Participants: Alarms
Arm/Group | Phase 2- Unblinded GE Portrait Monitoring
Number analyzed (Participants) | 73
Number analyzed (Alarms) | 73
Meaningful alarms | 60

3. Secondary Outcome: Phase 2 - Clinical Interventions to Meaningful Alarms
Description: Number of clinical interventions by the three categories of meaningful alarms (informative, important, and critical).
  An investigator will ask the relevant clinician (usually a nurse) to rate each alert as clinically meaningful or not. Specifically, clinicians will be asked to rate alerts as "critical," "important," "informative," or "false or distracting." The terms will intentionally not be further defined, thereby allowing caregivers to determine themselves the extent to which a given alert was helpful or not. Caregivers will be queried in person shortly after each alert, typically within 15 minutes. The thresholds, determined in the initial phase, will be set to generate an average of about 2 alerts per patient per day - and therefore will not be onerous for clinicians.
Time Frame: During postoperative 72 hours
Population: We analyzed 73 patients in the unblinded GE Portrait monitoring group, with a total of 73 alarms recorded. Among them, 41 patients experienced no alarms, while the remaining 32 patients accounted for all 73 alarms. Out of the 73 alarms, 60 alarms were categorized as informative, important, or critical by the responsible nurse.
Measure: Count of Units; unit: Meaningful alarms
Units Other Than Participants: Meaningful alarms
Arm/Group | Phase 2- Unblinded GE Portrait Monitoring
Number analyzed (Participants) | 73
Number analyzed (Meaningful alarms) | 60
Meaningful alarms
  Informative alarm: number analyzed (Meaningful alarms) | 30
  Informative alarm | 10
  Important alarm: number analyzed (Meaningful alarms) | 28
  Important alarm | 21
  Critical alarm: number analyzed (Meaningful alarms) | 2
  Critical alarm | 2

ADVERSE EVENTS:
Time Frame: During the first 72 postoperative hours
Groups:
- Phase 1 - Prospective Observational Cohort Study: Blinded GE Portrait Monitoring: Patients received continuous vital sign monitoring blinded to patients and clinicians.
  Phase 1 was a prospective cohort study and no randomization was done
- Phase 2- Randomized Trial: Unblinded GE Portrait Monitoring: Physician investigators monitored and evaluated continuous vital sign data 24 hours per day for patients assigned to unblinded GE Portrait monitoring.
Arm/Group | Phase 1 - Prospective Observational Cohort Study: Blinded GE Portrait Monitoring | Phase 2- Randomized Trial: Unblinded GE Portrait Monitoring | Phase 2- Randomized Trial: Blinded GE Portrait Monitoring
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/73 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/73 | 0/75
Other Adverse Events (participants affected / at risk) | 0/100 | 0/73 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/74/NCT05280574/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/74/NCT05280574/ICF_001.pdf